CLINICAL TRIAL: NCT01226030
Title: Dose Escalation and PK Study of M2ES in Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Protgen Ltd (Industry)
Responsible Party: Guodong Chang, Protgen Ltd
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-2008-2
Record Dates: First submitted 2010-10-09; First posted 2010-10-21 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-10

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- M2ES 7.5mg (Experimental): M2ES 7.5mg
  Interventions: Drug: M2ES 7.5mg
- M2ES 15mg (Experimental): M2ES 15mg
  Interventions: Drug: M2ES 15mg
- M2ES 30mg (Experimental): M2ES 30mg
  Interventions: Drug: M2ES 30mg
- M2ES 60mg (Experimental): M2ES 60mg
  Interventions: Drug: M2ES 60mg

INTERVENTIONS:
Drug: M2ES 7.5mg — M2ES 7.5mg
  Other Names: M2ES 7.5mg IV D1,8,15,22, every 28days a cycle.
  Arms: M2ES 7.5mg
Drug: M2ES 15mg — M2ES 15mg
  Other Names: M2ES 15mg IV D1,8,15,22, every 28days a cycle.
  Arms: M2ES 15mg
Drug: M2ES 30mg — M2ES 30mg
  Other Names: M2ES 30mg IV D1,8,15,22, every 28days a cycle.
  Arms: M2ES 30mg
Drug: M2ES 60mg — M2ES 60mg
  Other Names: M2ES 60mg IV D1,8,15,22, every 28days a cycle.
  Arms: M2ES 60mg

SUMMARY:
This study is dose-escalation open-label study to determine the MTD of M2ES in Subjects With Advanced Solid Tumors the recommended Phase II dose.The recommended dose and regimen of M2ES will be selected to perform the pharmacokinetic study profiles.

DETAILED DESCRIPTION:
This study is a Phase I dose-escalation open-label study to determine the MTD of M2ES in Subjects With Advanced Solid Tumors the recommended Phase II dose.The recommended dose and regimen of M2ES will be selected to perform the pharmacokinetic study profiles.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 60 years of age
2. patients had histologically or cytologically confirmed solid tumors that was refractory to standard therapy.
3. life expectancy of at least 3 months.
4. ECOGPS ≤ 1
5. Adequate hematologic, renal, and hepatic function was required as determined by the following: WBC ≥4×109/L, absolute neutrophil count ≥ 1.5×109/L, platelet count ≥100×109/L, hemoglobin ≥ 9g/dL, total bilirubin ≤1.5 upper limit of normal [ULN],AST ≤ 2.5 ULN, or ≤ 5 ULN if there was evidence of liver metastases; alkaline phosphatase ≤ 2.5 ULN, or ≤ 5 ULN if there was evidence of liver Metastases; creatinine clearance ≥50 mL/min.

Exclusion Criteria:

1. Pregnant and latent women, no contraception for women of childbearing age
2. Have taken other treatments
3. Be allergic to endostatin and other ingredient
4. Gastrointestinal Hemorrhage
5. Have Participated any clinical trail during the last 4 week
6. ECG: QTC ≥ 480 ms
7. patients had clinically apparent CNS disease ( primary brain tumors, tumor related apoplexy, CNS metastases, carcinomatous meningitis.)
8. Cardiovascular and mental disease
9. HIV-1 infected
10. HBV, HBV infected ,Hepatitis B surface antigen positive
11. Patients on therapeutic doses of heparin or antiplatelet agents.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-04 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerate dosage | 4 weeks
  The maxium tolerate dosage

SECONDARY OUTCOMES:
Pharmacokinetic (PK) behavior of M2ES in tumor subject | 4 week
  Pharmacokinetic (PK) behavior of different doses of M2ES in Subjects With Advanced Solid Tumors
The incidence rate of adverse event | 4 weeks
  The incidence rate of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, master, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China